CLINICAL TRIAL: NCT01861613
Title: Seroprevalence of Hepatitis B and Immune Response to Hepatitis B Vaccination in Chinese College Students
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hui Zhuang (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor-Investigator, Hui Zhuang, Professor, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HBV-001
Record Dates: First submitted 2013-05-19; First posted 2013-05-23 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis B; Immune Response; Seroprevalence
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B; halofantrine

ARMS (1):
- HBV vaccine (Experimental): HBV vaccine (Engerix-B, recombinant hepatitis B surface antigen, 20µg/mL/vial, GlaxoSmithKline, Belgium)
  Interventions: Biological: HBV vaccine (Engerix-B, recombinant hepatitis B surface antigen, 20µg/mL/vial, GlaxoSmithKline, Belgium)

INTERVENTIONS:
Biological: HBV vaccine (Engerix-B, recombinant hepatitis B surface antigen, 20µg/mL/vial, GlaxoSmithKline, Belgium)

SUMMARY:
At present, children less than 15 y of age have been regarded as a key group for hepatitis B immunization in China. However, there is not yet special immunization strategy for population above 15 y of age. In this study, we investigated the seroprevalence of hepatitis B and immune response to HB vaccine among Chinese college students to uncover the need on universal mass vaccination or booster immunization only for students with HBV vaccination history against hepatitis B in Chinese college students to inform decision making.

ELIGIBILITY:
Inclusion Criteria:

* Male and female freshmen in one college in Liuzhou city of Guangxi Zhuang Autonomous Region

Exclusion Criteria for vaccination study:

* acute illness
* immunocompromised conditions
* renal insufficiency
* pregnancy
* allergic history to HB vaccine or yeast
* positive for any of HBsAg, anti-HBs or anti-HBc

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2040 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Anti-HBs immune response in participants negative for HB sAg, anti-HBs and anti-HBc | Anti-HBs was assayed at Month 7

SECONDARY OUTCOMES:
Seroprevalence for HBsAg, anti-HBs and anti-HBc in Chinese college students | seroprevalence at baseline
Anti-HBs immune response in participants negative for HBsAg, anti-HBs and anti-HBc | Anti-HBs immune response at Month 1
Anti-HBs immune response in participants negative for HBsAg, anti-HBs and anti-HBc | Anti-HBs immune response at Month 6
Anti-HBs immune response in participants negative for HBsAg, anti-HBs and anti-HBc | Anti-HBs immune response at Month 20

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Centers for Disease Control and Prevention, Nanning, Guangxi, China